CLINICAL TRIAL: NCT01003145
Title: A Clinical Study to Assess the Immunogenicity and Safety of Influenza Virus Vaccine, AdimFlu-S (A/H1N1), in Healthy Volunteers
Brief Title: Immunogenicity and Safety of Influenza Virus Vaccine, AdimFlu-S (A/H1N1), in Adults and Elders
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Adimmune Corporation (Industry)
Responsible Party: Jeffrey Chen / Vice President, Adimmune Corporation
Allocation: Randomized | Masking: None | Purpose: Prevention
Other Study IDs: FLU09001
Record Dates: First submitted 2009-10-27; First posted 2009-10-28 (Estimated); Last update posted 2012-01-20 (Estimated); Status verified 2012-01

CONDITIONS: Influenza
Keywords: Influenza; vaccine; Immunogenicity
MeSH Terms: conditions — Influenza, Human

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- H1N1 vaccine of 15 μg HA on Day 0 (Experimental): 15 μg HA (0.5 mL) per injection, 1 injection
  50 adults (aged 18~60 years) were assigned to receive one injection of H1N1 vaccine
  Interventions: Biological: Influenza A (H1N1) 2009 monovalent vaccine, inactivated
- H1N1 vaccine of 15 μg HA on Day 0 and 21 (Experimental): 15 μg HA (0.5 mL) per injection, 2 injections
  50 adults (aged 18~60 years) and 50 elders (aged over 60 years) were assigned to receive two injections of H1N1 vaccine 3 weeks apart
  Interventions: Biological: Influenza A (H1N1) 2009 monovalent vaccine, inactivated
- H1N1 vaccine of 30 μg HA on Day 0 and 21 (Experimental): 30 μg HA (1 mL) per injection, 2 injections
  50 adults (aged 18~60 years) and 50 elders (aged over 60 years) were assigned to receive two injections of H1N1 vaccine 3 weeks apart
  Interventions: Biological: Influenza A (H1N1) 2009 monovalent vaccine, inactivated

INTERVENTIONS:
Biological: Influenza A (H1N1) 2009 monovalent vaccine, inactivated
  Other Names: AdimFlu-S (A/H1N1)

SUMMARY:
This was a randomized, laboratory-blinded study in healthy male and non-pregnant female designed to investigate the safety, reactogenicity, and immunogenicity of an inactivated influenza H1N1 vaccine (AdimFlu-S). In the adult cohort, all volunteers were randomized in a 1:1:1 ratio to receive 2 injections of AdimFlu-S (A/H1N1) 15 mcg HA at 3 weeks apart, 2 injections of AdimFlu-S (A/H1N1) 30 mcg HA at 3 weeks apart or 1 injection of AdimFlu-S (A/H1N1) 15 mcg HA. In the elders cohort, all volunteers were randomized in a 1:1 ratio to receive 2 injections of AdimFlu-S (A/H1N1) 15 mcg HA at 3 weeks apart or 2 injections of AdimFlu-S (A/H1N1) 30 mcg HA at 3 weeks apart.

Following immunization, safety was measured by assessment of adverse events for 6 weeks following the first vaccination, serious adverse events and new-onset chronic medical conditions through 7 months post first vaccination; and reactogenicity to the vaccines for 7 days following each vaccination. Immunogenicity testing included hemagglutinin inhibition (HAI) testing on serum obtained before first vaccination, and three and six weeks after first vaccination.

ELIGIBILITY:
Inclusion Criteria:

* Males or non-pregnant females and age ≧ 18 years;
* Willing and able to adhere to visiting schedules and all study requirements;
* In good physical health on the basis of medical history, physical examination;
* Subject should read and sign the study-specific informed consent.

Exclusion Criteria:

* Subject ever received influenza vaccine within the previous 6 months;
* History of hypersensitivity to eggs or egg protein or similar pharmacological effects to study medication (AdimFlu-S (A/H1N1));
* Personal or family history of Guillain-Barré Syndrome;
* An acute febrile illness within the last 72 hours prior to vaccination;
* Subjects, with bleeding or any coagulation disorder, who receive anticoagulants in the preceding 3 weeks, thus posing a contraindication for intramuscular injection;
* Subjects with influenza-like illness as defined by the presence of fever (temperature ≧38.5℃) and at least two of the following four symptoms: headache, muscle/joint aches and pains (e.g. myalgia/arthralgia), sore throat and cough;
* Female subjects who are pregnant, lactating or likely to become pregnant during the study. Women of childbearing potential who disagree to use an acceptable method of contraception (e.g., hormonal contraceptives, IUD, barrier device or abstinence) throughout the study;
* Treatment with an investigational drug or device, or participation in a clinical study, within 3 months before consent;
* Immunodeficiency, immunosuppressive or household contact with immunosuppression;
* History of wheezing or have been using bronchodilator within 3 months prior to study vaccination;
* Receipt of live virus vaccine within 1 month prior to study vaccination or expected receipt within 2 months after first study vaccination;
* Receipt of any inactivated vaccine within 2 weeks prior to study vaccination or expected receipt of vaccination within 3 weeks after the immunogenicity evaluation period;
* Receipt of any blood products, including immunoglobulin in the prior 3 months;
* Underlying condition, in the investigator's opinion, that may be inappropriate for vaccination;
* Significant chronic illness for which inactivated influenza vaccine is recommended or commonly used.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 292 (Actual)
Dates: Start 2009-09; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
The primary immunogenicity objective is to assess the antibody response following a single dose of study vaccine, stratified by age of recipient, when administered at the 15 or 30 μg HA doses.
The primary safety objective of this study is to assess the safety of the study vaccine when administered at the 15 or 30 μg dose.

SECONDARY OUTCOMES:
The secondary immunogenicity objective is to assess the antibody response following 2 doses of study vaccine, stratified by age of recipient, when administered at the 15 or 30 μg HA doses.

CONTACTS AND LOCATIONS:
Overall Officials: Szu Min Hsieh, Principal Investigator — National Taiwan University Hospital; Feng Yee Chang, Principal Investigator — Tri-Service General Hospital; Yung Ching Liu, Principal Investigator — Taipei Medical University Wang Fang Hospital
Locations (3):
- Taiwan (3):
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Wang Fang Hospital, Taipei
  - Tri-Service General Hospital, Taipei

REFERENCES:
- [Derived] Kung HC, Huang KC, Kao TM, Lee YC, Chang FY, Wang NC, Liu YC, Lee WS, Liu HJ, Chen CI, Chen CH, Huang LM, Hsieh SM. A clinical study to assess the immunogenicity and safety of a monovalent 2009 influenza A (H1N1) vaccine in an area with low-level epidemics of pandemic influenza. Vaccine. 2010 Oct 21;28(45):7337-43. doi: 10.1016/j.vaccine.2010.08.073. Epub 2010 Sep 17. PMID 20817013
- [Derived] Kao TM, Hsieh SM, Kung HC, Lee YC, Huang KC, Huang LM, Chang FY, Wang NC, Liu YC, Lee WS, Liu HE, Chen CI, Chen CH. Immune response of single dose vaccination against 2009 pandemic influenza A (H1N1) in the Taiwanese elderly. Vaccine. 2010 Aug 31;28(38):6159-63. doi: 10.1016/j.vaccine.2010.07.026. Epub 2010 Jul 24. PMID 20659517